CLINICAL TRIAL: NCT05239455
Title: An In Vivo 24-Hour Recovery Study of Leukoreduced RBCs After Automated Separation of Whole Blood by the Reveos System and Storage for 42 Days
Brief Title: An In Vivo 24-Hour Recovery Study of Whole Blood by the Reveos System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Terumo BCT (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CTS-5085
Record Dates: First submitted 2022-01-03; First posted 2022-02-14 (Actual); Results first posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2023-04

CONDITIONS: Device Validation of In-vivo Performance
Keywords: Reveos; Reveos Device; Reveos System; Red Blood Cell Storage; Whole Blood Processing; In-vivo 24-hour red blood cell recovery; Reveos System Manager; Reveos SELECT Set US; Reveos In Vivo US

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Healthy adult participants (Experimental): Performance criteria will be evaluated in healthy adult participants, who receive radiolabeled, autologous infusions of LR-RBC components after being stored for 42 days at 1-6°C.
  Interventions: Device: Reveos® Automated Blood Processing System

INTERVENTIONS:
Device: Reveos® Automated Blood Processing System — This is a non-interventional study, observing the in vivo performance of LR-RBC units derived from WB processed with the Reveos System.

SUMMARY:
This is an in vivo 24-hour recovery study of leukoreduced red blood cells (RBCs) after automated separation of whole blood by the Reveos Automated Blood Processing System and storage for 42 days.

DETAILED DESCRIPTION:
The Reveos® Automated Blood Processing System (Reveos system) is an automated whole blood processing system, not cleared for use in the United States. The Reveos System has been available outside the United States since 2012 and is seeking United States Food and Drug Administration (FDA) 510(k) clearance as an automated whole blood processor. The Reveos System is an integrated manufacturing system that processes whole blood (WB) units into blood components and is designed to minimize manual blood processing variables resulting from processing time, product and procedural variability. The Reveos System can simultaneously process up to 4 whole blood units into 4 RBC units, 4 leukoreduced plasma units, and 4 interim platelet units (IPU). The CPD/AS-5 RBC product is leukoreduced and may be stored up to 42 days.

Terumo BCT is seeking 510(k) clearance from FDA/CBER for the Reveos® Automated Blood Processing System (Reveos System). The proposed study will provide validation on the in vivo performance of LR-RBC units derived from WB processed with the Reveos System. The results will provide data as to whether the Reveos System produced LR-RBC can maintain required levels of 24-hour in vivo recovery that meet FDA criteria for RBC.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers, of either gender
2. Age 18 years or older.
3. Normal health status as per AABB criteria for healthy donor.
4. Able to commit to the study schedule.
5. Meets the inclusion criteria defined by the Blood Center for whole blood donor. These criteria are based on FDA Regulations and AABB standards. Note: Participants who are deferred from volunteer community donations because of travel restrictions, piercings, tattoos or other reasons by PI approval may participate in the study, as products are re-transfused to the autologous donor.
6. Participants of childbearing potential (either male or female) must agree to use medically acceptable method of contraception throughout of the study.
7. Females of childbearing potential must be willing to take a pregnancy test prior to WB donation and infusion of radiolabeled RBCs.
8. Signed and dated informed consent form.

Exclusion Criteria:

1. Pregnant or nursing females.
2. Serum ferritin <12 ng/mL
3. Has previously completed this study with evaluable data points.
4. Participation currently, or within the past 30 days, in another investigational trial that would potentially interfere with the analysis of this investigation (eg, pharmaceutical).
5. As determined by the Investigator

   1. Has been diagnosed with a blood disorder(s) affecting RBC characteristics (eg, G- 6PD).
   2. Reported history of RBC autoantibodies/autoimmune hemolytic anemia, RBC alloantibodies.
   3. Clinically significant acute or chronic disease
   4. Reported history of known hypersensitivity to technetium or chromium.
   5. Treatment with any medication as specified in site deferral list (based on AABB medication deferral list for blood donors).
6. Other unspecified reasons that, in the opinion of the investigator make the subject unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Cancelas, MD, PhD, Principal Investigator — Hoxworth Blood Center, University of Cincinnati; Moritz Stolla, MD, PhD, Principal Investigator — Bloodworks Northwest Research Institute; James Kelley, MD, PhD, Study Chair — Terumo BCT
Locations (2):
- United States (2):
  - Hoxworth Blood Center, University of Cincinnati, Cincinnati, Ohio
  - Bloodworks Northwest Research Institute, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A donor is considered an "enrolled" participant upon giving informed consent for study participation; this timepoint represents the beginning of a participant's involvement in the study.
Pre-assignment Details: 37 participants signed consent and there were 4 screen fails.
Period: Overall Study
Arm/Group | Healthy Adult Participants
Started | 33
Completed | 26
Not Completed | 7
Not completed — Adverse Event | 1
Not completed — Sponsor Decision | 5
Not completed — Incomplete Blood Collection | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Population includes all participants that met the eligibility criteria.
Arm/Group | Healthy Adult Participants
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (17.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 28
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 33
Height [Mean (Standard Deviation); unit: inches] | 69.15 (4.617)
Weight [Mean (Standard Deviation); unit: lbs] | 192.6 (37.47)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Success of RBC's in Vivo Recovery After 42-day Storage
Description: The primary outcome of this study is to measure mean 24-hour, post-transfusion, in vivo RBC recovery percentage after LR-RBCs derived from WB and processed with the Reveos System have been stored for 42-days at 1-6°C.
  The 3 parts of FDA's RBC recovery criteria that must be met (below) are presented in Primary Outcome 1 and Primary Outcome 2. The derivation of the sample size was based on the level of precision attained with 24 subjects relative to the 1st part of the criteria.
  1. The one-sided 95% lower confidence limit for the population proportion of success is greater than 70% where success of a unit is defined as the RBC in vivo 24-hour percentage recovery
     ≥ 75% [Allows for low recoveries (<75%) in 2/20 or 3/24 volunteers] - Primary Outcome 1
  2. The sample mean of percent recovery ≥ 75% - Primary Outcome 2
  3. The sample standard deviation of in vivo 24-hour RBC recovery ≤ 9% - Primary Outcome 2
Time Frame: 43 days
Population: The Evaluable Analysis Population includes all participants who completed all study visits per the CIP with a valid 24-hour recovery endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Adult Participants
Number analyzed (Participants) | 26
Participants | 23
Statistical Analysis 1: Comparison: Healthy Adult Participants; The comparison is to the FDA requirements for in vivo 24-hour recovery of LR-RBC; Test type: Other — The FDA requires one-sided 95% lower confidence limit for the population proportion of success is greater than 70% where success of a unit is defined as the RBC in vivo 24-hour percentage recovery ≥ 75%. Allows for low recoveries (<75%) in 2/20 or 3/24 volunteers; 95% Confidence Interval = 88.5, 95% CI 1-sided [lower limit 72.81] — A one-sided confidence interval for the proportion of successes was determined using the Clopper-Pearson exact method for a 95% confidence interval; Proportion of successes greater than 70% where success of a unit is defined as the RBC in vivo 24-hour percentage recovery ≥ 75% was calculated

2. Primary Outcome: Mean 24-hour, Post-transfusion, in Vivo RBC Recovery Percentage After 42-day Storage
Description: as for outcome 1
Time Frame: 43 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % 24-hr RBC Recovery
Arm/Group | Healthy Adult Participants
Number analyzed (Participants) | 26
% 24-hr RBC Recovery | 83 (9)
Statistical Analysis 1: Comparison: Healthy Adult Participants; The comparison is to the FDA requirements for in vivo 24-hour recovery of LR-RBC; Test type: Other — The FDA criteria requires LR-RBC mean 24-hour recovery ≥ 75% with standard deviation (SD) ≤ 9%; Mean and standard deviation were calculated

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of signing the informed consent through study completion. Adverse event assessments occurred at Day 0, Day 42, and Day 43. There was no long term follow-up.
Description: Only procedure emergent AEs (PEAEs) were included in the safety evaluation. Collection of PEAEs began at the time of the first exposure to Reveos Blood Bag set and continued throughout the entire study until study exit or observed related AEs were resolved. Starting with the first baseline procedure, any new event/experience that was not present at baseline, or worsening of an event present at baseline, was considered an AE.
Arm/Group | Healthy Adult Participants
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 2/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Healthy Adult Participants (N=33)
Vessel puncture site bruise (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Available upon request.

DOCUMENTS (2):
  • Study Protocol (2022-03-11): https://cdn.clinicaltrials.gov/large-docs/55/NCT05239455/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/55/NCT05239455/SAP_001.pdf